CLINICAL TRIAL: NCT03269188
Title: Incidence and Associated Factors of Persistent Postoperative Incision Scar Pain Following C/s in Mulago Hospital
Acronym: PPOPinC/S
Status: Completed | Type: Observational
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: Persistent pain in C/S
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
prospective cohort study of women who underwent caesarean section in mulago hospital. followed up for 2 months and assessed for development of persistent post operative pain at the incision site and its effect on quality of life. incidence of persistent postoperative pain and associated factors determined.

DETAILED DESCRIPTION:
prospective cohort study of 277 women who underwent caesarean section in mulago hospital. demographic, medical history, intraoperative, postoperative details, and perioperative levels of pain collected. followed up by telephone interviews for 2 months and assessed for development of persistent post operative pain at the incision site and its effect on quality of life. incidence of persistent postoperative pain and associated factors determined.

ELIGIBILITY:
Inclusion Criteria:

- ASA I, II, and III.

* patient who has given informed consent.

Exclusion Criteria:

* patients who have no telephone contact

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: women scheduled to undergo both elective and emergency caesarean section in the obstetric theatres of mulago national referral hospital during the study period and meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2016-10-10 (Actual); Study Completion 2016-10-27 (Actual)

PRIMARY OUTCOMES:
persistent postoperative pain at caesarean section incision scar site. | 2 months.
  participant report pain at site of caesarean section incision site scar at 2 months after caesarean section.